CLINICAL TRIAL: NCT03076099
Title: Effects of Dexmedetomidine on Post-operative Blood Pressure in Patients Undergoing Brain Arteriovenous Malformation Embolization
Brief Title: Dexmedetomidine on Post-operative Blood Pressure in Bain Arteriovenous Malformation Embolization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nan Jiang (Other)
Responsible Party: Sponsor-Investigator, Nan Jiang, associate professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NJiang2016-001
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia
Keywords: Dexmedetomidine; brain arteriovenous malformation; embolization; post-operative hypertension
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: two parallel groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: this investigation is a triple mask study. The patiens, the care providers and Outcome Assessor will not allowed to know the grouping information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine was administered intravenously when tracheal extubation, 1.2μg/kg Dexmedetomidine was mixed with 100 ml normal saline and maintained 4 hours constantly.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Normal Saline was administered intravenously when tracheal extubation,equal volume of normal saline was mixed with 100 ml normal saline and maintained 4 hours constantly.
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — 1.2 μg/kg Dexmedetomidine was administered intravenously constantly after tracheal extubation.
  Other Names: DEX
  Arms: Dexmedetomidine
Other: normal saline — equal volume of normal saline was administered intravenously constantly after tracheal extubation.
  Other Names: NS
  Arms: Control group

SUMMARY:
Aim of this trial is to study the effect of Dexmedetomidine on post-operative blood pressure in patients undergoing brain arteriovenous malformation embolization. The patients were randomized allocated to either Dexmedetomidine group or Control group. Patients in Dexmedetomidine group will receive intravenous Dexmedetomidine while the control group will receive normal saline. Post-operative anti-hypertensive drug, Visual analogue score,post-operative analgesics consumption, Quality of Recovery score, Ramsay score, and adverse events were recorded.

DETAILED DESCRIPTION:
Aim of this trial is to study the effect of Dexmedetomidine on post-operative blood pressure in patients undergoing brain arteriovenous malformation embolization. The patients were randomized allocated to either Dexmedetomidine group or Control group according to a random number. Patients in Dexmedetomidine group will receive intravenous Dexmedetomidine while the control group will receive normal saline. Post-operative anti-hypertensive drug, Visual analogue score,post-operative analgesics consumption, Quality of Recovery score-15 items, Ramsay score, and adverse events were recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing brain arteriovenous malformation embolization in the fist affiliated hospital, Sun Yat-sen University, aged 18-65 years, available to chat with,and the tracheal tube was extubated after surgery immediately.

Exclusion Criteria:

* abuse anesthetic analgesics and sedative drugs, or allergic to Dexmedetomidine or other anesthetics, hypotension or bradycardia before surgery, severe pulmonary disease with saturation of pulse oximetry less than 90% before surgery, or patients refused to attend in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
urapidil consumption | the end of the 6th hour after tracheal extubation
  urapidil consumption was recorded by nurses every hour

SECONDARY OUTCOMES:
urapidil consumption on POD1 | the total consumption of urapidil on post-operative day 1.
  urapidil consumption was recorded by nurses every hour
urapidil consumption on POD2 | the total consumption of urapidil on post-operative day 2.
  urapidil consumption was recorded by nurses every hour
Visual Analogue score | the end of the 6th hour after tracheal extubation
  visual analogue score was measured by visual analogue scale
Visual Analogue score at 24th hour | the end of the 24th hour after tracheal extubation
  visual analogue score was measured by visual analogue scale
Visual Analogue score at 48th hour | the end of the 48th hour after tracheal extubation
  visual analogue score was measured by visual analogue scale
Quality of Recovery Score | the end of the 6th hour after tracheal extubation
  Quality of Recovery Score was measured by a 15-item quality of recovery scale
Quality of Recovery Score at 24th hour | the end of the 24th hour after tracheal extubation
  Quality of Recovery Score was measured by a 15-item quality of recovery scale
Quality of Recovery Score at 48th hour | the end of the 48th hour after tracheal extubation
  Quality of Recovery Score was measured by a 15-item quality of recovery scale
Analgesics consumption | the end of the 6th hour after tracheal extubation
  Analgesics consumption was recorded by nurse every hour
Analgesics consumption on POD1 | the total consumption of urapidil on post-operative day 1.
  Analgesics consumption was recorded by nurse every hour
Analgesics consumption on POD2 | the total consumption of urapidil on post-operative day 2.
  Analgesics consumption was recorded by nurse every hour
Bradycardia | the end of the 6th hour after tracheal extubation
  a heart rate of lower than 50 beats per minute was identified as bradycardia, frequency of bradycardia was recorded by nurse
Bradycardia at 24th hour | the end of the 24th hour after tracheal extubation
  a heart rate of lower than 50 beats per minute was identified as bradycardia, frequency of bradycardia was recorded by nurse
Bradycardia at 48th hour | the end of the 48th hour after tracheal extubation
  a heart rate of lower than 50 beats per minute was identified as bradycardia, frequency of bradycardia was recorded by nurse
PONV | the end of the 6th hour after tracheal extubation
  post-operative nausea and vomiting (PONV) was recorded by nurse
PONV at 24th hour | the end of the 24th hour after tracheal extubation
  post-operative nausea and vomiting (PONV) was recorded by nurse
PONV at 48th hour | the end of the 48th hour after tracheal extubation
  post-operative nausea and vomiting (PONV) was recorded by nurse

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Sun Yetsen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
the IPD will not be shared with others, since following investigations based on this trial is about to start.